CLINICAL TRIAL: NCT06457139
Title: Preventing Type 2 Diabetes Mellitus After Gestational Diabetes Mellitus With Immediate Postpartum Screening
Brief Title: Preventing T2DM After GDM With Immediate Postpartum Screening
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Gianna Wilkie, Assistant Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: STUDY00001870
Record Dates: First submitted 2024-06-06; First posted 2024-06-13 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Gestational Diabetes; Type 2 Diabetes
Keywords: diabetes
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Glucose Tolerance Test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Postpartum GDM Screening (Experimental): Subjects who are randomly assigned to this condition will be screened for GDM with the recommended 2-hour glucose tolerance test during their postpartum hospitalization.
  Interventions: Diagnostic Test: Glucose tolerance test (2 hour)
- Standard of Care Postpartum Screening (Active Comparator): Subjects randomized to the comparison condition will receive the usual standard of care. The standard of care will consist of screening with a 2 hour glucose tolerance test at 6-12 weeks postpartum.
  Interventions: Other: Active Comparator

INTERVENTIONS:
Diagnostic Test: Glucose tolerance test (2 hour) — Early testing with the 2 hour glucose tolerance test will occur during their inpatient postpartum hospitalization.
  Arms: Early Postpartum GDM Screening
Other: Active Comparator — Subjects randomized to the comparison condition will receive the usual standard of care. The standard of care will consist of administration of educational materials adapted from the American Diabetes Association that discusses healthy lifestyle behaviors and the increased risks of developing T2DM after a pregnancy complicated by GDM.
  Arms: Standard of Care Postpartum Screening

SUMMARY:
The overall goal of this proposal is to create and test an implementation protocol for in-hospital immediate postpartum diabetes screening for postpartum patients with pregnancies affected by GDM.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) affects 6 to 8% of U.S. pregnancies annually and upwards of 1 in every 8 pregnancies worldwide. Pregnant individuals with GDM have higher rates of hypertensive disorders of pregnancy, cesarean delivery, and maternal mortality as compared to those without GDM. While GDM frequently resolves after delivery, up to 70% of patients will develop type 2 diabetes mellitus (T2DM) later in life10 and one third will develop subsequent diabetes or impaired glucose metabolism at the time of postpartum screening.

While postpartum screening is recommended by the American College of Obstetricians and Gynecologists (ACOG) and the American Diabetes Association (ADA) between 4-12 weeks postpartum for all patients with GDM in pregnancy, nearly 40% of patients do not attend a postpartum visit. Attendance is even lower among populations with limited resources, contributing to health disparities.

To address this issue, immediate in-hospital postpartum glucose tolerance testing has been evaluated and found to yield diagnostic values comparable to postpartum screening with the advantage of ~100% adherence. However, 2 challenges remain: currently there is a lack of widespread clinical implementation of in-hospital immediate postpartum diabetes screening.

Therefore, the overall goal of this proposal is to randomize patients to early screening during their postpartum hospitalization versus at their 6 week postpartum visit (current standard of care).

ELIGIBILITY:
Inclusion Criteria:

* pregnancy complicated by GDM as diagnosed with traditional two step testing in the third trimester according to Carpenter-Coustan Criteria
* receiving prenatal care at UMASS Memorial and plans to deliver at UMASS Memorial
* able and willing to provide informed consent
* ability to complete immediate in hospital postpartum glucose testing
* have evidence of impaired glucose metabolism defined as fasting glucose value of ≥126 mg/dL or 2-hour glucose value of ≥200 mg/dL

Exclusion Criteria:

* known diagnosis of pre-existing pre-gestational diabetes in pregnancy
* inability to complete oral glucose tolerance test (e.g. gastric bypass surgery history, gastric dumping syndrome history, vomiting of oral glucose tolerance test) in pregnancy or immediately postpartum
* systemic steroid use

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Detection of Type 2 Diabetes Mellitus | At time of postpartum screening (postpartum day 1 or 6 week postpartum visit pending randomization arm)
  Detection of Type 2 Diabetes Mellitus by 2 hour oral glucose tolerance test
Glycemic Outcomes--Hemoglobin A1c | at time of postpartum screening (postpartum day 1 or 6 week postpartum visit pending randomization arm)
  Serum blood measurement of hemoglobin A1c

SECONDARY OUTCOMES:
Patient Satisfaction | At postpartum visit (6 weeks after delivery)
  Participant satisfaction will be assessed using the validated survey, the Patient Satisfaction Survey. The survey was developed in 1979 and has been used to assess patient satisfaction with research participation based on 8 simple questions. It has not been used in a randomized trial in an obstetric population but has been validated in other clinical populations
Patient Recruitment | at time of randomization (postpartum day 1)
  The investigators will examine the total number of subjects that were approached and the reasons for ineligibility and non-participation.
Patient Retention | At postpartum visit (6 weeks after delivery)
  The investigators will record reasons for failure to complete in hospital diabetes screening and treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gianna Wilkie, MD, Principal Investigator — UMASS Memorial Healthcare
Locations (1):
- University of Massachusetts Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Werner EF, Has P, Rouse D, Clark MA. Two-day postpartum compared with 4- to 12-week postpartum glucose tolerance testing for women with gestational diabetes. Am J Obstet Gynecol. 2020 Sep;223(3):439.e1-439.e7. doi: 10.1016/j.ajog.2020.05.036. Epub 2020 May 26. PMID 32470456
- [Background] Waters TP, Kim SY, Werner E, Dinglas C, Carter EB, Patel R, Sharma AJ, Catalano P. Should women with gestational diabetes be screened at delivery hospitalization for type 2 diabetes? Am J Obstet Gynecol. 2020 Jan;222(1):73.e1-73.e11. doi: 10.1016/j.ajog.2019.07.035. Epub 2019 Jul 24. PMID 31351065
- [Background] Dinglas C, Muscat J, Heo H, Islam S, Vintzileos A. Immediate Postpartum Glucose Tolerance Testing in Women with Gestational Diabetes: A Pilot Study. Am J Perinatol. 2017 Oct;34(12):1264-1270. doi: 10.1055/s-0037-1606620. Epub 2017 Sep 14. No abstract available. PMID 28910846
- [Background] Ratner RE, Christophi CA, Metzger BE, Dabelea D, Bennett PH, Pi-Sunyer X, Fowler S, Kahn SE; Diabetes Prevention Program Research Group. Prevention of diabetes in women with a history of gestational diabetes: effects of metformin and lifestyle interventions. J Clin Endocrinol Metab. 2008 Dec;93(12):4774-9. doi: 10.1210/jc.2008-0772. Epub 2008 Sep 30. PMID 18826999
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527